CLINICAL TRIAL: NCT03882970
Title: A Randomized, Phase 3, Open-Label Trial Comparing the Effect of LY3298176 Versus Titrated Insulin Degludec on Glycemic Control in Patients With Type 2 Diabetes
Brief Title: A Study of Tirzepatide (LY3298176) Versus Insulin Degludec in Participants With Type 2 Diabetes
Acronym: SURPASS-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16997; I8F-MC-GPGH (Other: Eli Lilly and Company); 2018-003422-84 (EudraCT Number)
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide; insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 5 mg Tirzepatide (Experimental): 5 milligrams (mg) tirzepatide administered subcutaneously (SC) once a week.
  Interventions: Drug: Tirzepatide
- 10 mg Tirzepatide (Experimental): 10 mg tirzepatide administered SC once a week.
  Interventions: Drug: Tirzepatide
- 15 mg Tirzepatide (Experimental): 15 mg tirzepatide administered SC once a week.
  Interventions: Drug: Tirzepatide
- Insulin Degludec (Active Comparator): Insulin degludec administered SC once a day.
  Interventions: Drug: Insulin Degludec

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 10 mg Tirzepatide; 15 mg Tirzepatide; 5 mg Tirzepatide
Drug: Insulin Degludec — Administered SC
  Arms: Insulin Degludec

SUMMARY:
The purpose of this study is to compare the effect of the study drug tirzepatide to insulin degludec on blood sugar levels in participants with type 2 diabetes. The study will last about 67 weeks and may include up to 22 visits.

ELIGIBILITY:
Inclusion Criteria:

* Participants must:

  * Have been diagnosed with type 2 diabetes mellitus (T2DM)
  * Have HbA1c between ≥7.0% and ≤10.5%
  * Be on stable treatment with unchanged dose of metformin or metformin plus an SGLT-2 inhibitor for at least 3 months before screening
  * Be of stable weight (± 5%) for at least 3 months before screening
  * Have a BMI ≥25 kilograms per meter squared (kg/m2) at screening

Exclusion Criteria:

* Participants must not:

  * Have type 1 diabetes mellitus
  * Have had chronic or acute pancreatitis any time prior to study entry
  * Have proliferative diabetic retinopathy or diabetic maculopathy or nonproliferative diabetic retinopathy requiring acute treatment
  * Have disorders associated with slowed emptying of the stomach, or have had any stomach surgeries for the purpose of weight loss
  * Have acute or chronic hepatitis, signs and symptoms of any other liver disease, or blood alanine transaminase (ALT) enzyme level >3.0 times the upper limit of normal (ULN) for the reference range, as determined by the central laboratory. Participants with nonalcoholic fatty liver disease (NAFLD) are eligible for participation in this trial only if their ALT level is ≤3.0 the ULN for the reference range
  * Have an estimated glomerular filtration rate <45 mL/minute/1.73 m2 (or lower than the country specific threshold for using the protocol required dose of metformin per local label)
  * Have had a heart attack, stroke, or hospitalization for congestive heart failure in the past 2 months
  * Have a personal or family history of medullary thyroid carcinoma or personal history of multiple endocrine neoplasia syndrome type 2
  * Have been taking any other diabetes medicines other than metformin, or metformin plus an SGLT-2 inhibitor during the last 3 months
  * Have been taking weight loss drugs, including over-the-counter medications during the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1444 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2021-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (121):
- United States (32):
  - Arkansas Clinical Research, Little Rock, Arkansas
  - Valley Research, Fresno, California
  - National Research Institute, Huntington Park, California
  - National Research Institute, Los Angeles, California
  - Catalina Research Institute, LLC, Montclair, California
  - Valley Clinical Trials, Inc., Northridge, California
  - National Research Institute, Panorama City, California
  - Encompass Clinical Research, Spring Valley, California
  - University Clinical Investigators, Inc., Tustin, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - East Coast Clinical Research, Jacksonville, Florida
  - East Coast Institute For Research, Jacksonville, Florida
  - Bayside Clinical Research, LLC, New Port Richey, Florida
  - East Coast Institute For Research, Macon, Georgia
  - Sky Clinical Research Network, Union City, Georgia
  - Elite Clinical Trials LLLP, Blackfoot, Idaho
  - Humphreys Diabetes Center, Boise, Idaho
  - Rocky Mountain Diabetes and Osteoporosis Center, Idaho Falls, Idaho
  - Springfield Diabetes & Endocrine Center, Springfield, Illinois
  - Crescent City Clinical Research, Metairie, Louisiana
  - Endocrine and Metabolic Consultants, Rockville, Maryland
  - Troy Internal Medicine, PC, Troy, Michigan
  - International Diabetes Center, Minneapolis, Minnesota
  - Clinical Research Professionals, Chesterfield, Missouri
  - Palm Research Center, Las Vegas, Nevada
  - Aventiv Research, Columbus, Ohio
  - The Corvallis Clinic P.C., Corvallis, Oregon
  - Heritage Valley Medical Group, Inc., Beaver, Pennsylvania
  - Detweiler Family Medicine, Lansdale, Pennsylvania
  - Office of Dr. Osvaldo Brusco, Corpus Christi, Texas
  - Consano Clinical Research, Shavano Park, Texas
- Argentina (9):
  - Mautalen Salud e Investigación - Servicio de Endocrinología, CABA, Buenos Aires
  - Investigaciones Medicas IMOBA S.R.L., Caba, Buenos Aires
  - CEDIC-Centro de Investigaciones Clinicas, Caba, Buenos Aires
  - Centro de Investigacion y Prevencion Cardiovascular (CIPREC), Ciudad Autonoma de, Buenos Aires
  - CIPADI, Godoy Cruz, Mendoza Province
  - AXISMED SRL - Bioclinica Research Network, Buenos Aires
  - Centro Médico Viamonte, Ciudad Autonoma de Buenos Aire
  - Instituto Centenario, Ciudad Autonoma de Buenos Aire
  - CENUDIAB, Ciudad Autonoma de Buenos Aire
- Austria (4):
  - Landesklinikum Korneuburg-Stockerau, Standort Stockerau, Stockerau, Lower Austria
  - Universitätsklinikum Graz, Graz, Styria
  - Universitätsklinikum Salzburg, Salzburg
  - KA Rudolfstiftung, Vienna
- Greece (10):
  - Iatriko Palaiou Falirou, Medical Center, Palaió Fáliro, Athens
  - Laiko General Hospital of Athens, Ampelokipoi, Attica
  - Gen Hospital of Athens G Gennimatas, Athens, Attica
  - General Hospital of Thessaloniki Papageorgiou, N. Efkarpia, Thessaloniki
  - Thermi Clinic, Thermi, Thessaloniki
  - Athens Euroclinic, Athens
  - University General Hospital of Larissa, Larissa
  - AHEPA Hospital, Thessaloniki
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki
  - Euromedica - General Clinic of Thessaloniki, Thessaloniki
- Hungary (8):
  - Kenezy Gyula Korhaz es Rendelointezet, Debrecen, Hajdú-Bihar
  - Szent Margit Rendelointezet, Budapest
  - ClinDiab Kft., Budapest
  - XIII.ker Onkormanyzat Egeszsegugyi Szolgalat, Budapest
  - Strazsahegy Medicina Bt., Budapest
  - TRANTOR 99 Bt., Budapest
  - Kanizsai Dorottya Korhaz, Nagykanizsa
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- Italy (6):
  - Azienda ospedaliero-universitaria Mater Domini, Germaneto, Catanzaro
  - Policlinico Univ. Agostino Gemelli, Rome, Lazio
  - Centro Cardiologico Monzino, IRCCS, Milan, MI
  - Azienda Ospedaliera Policlinico Consorziale, Bari
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Ospedale Santa Maria Goretti, Latina
- Poland (8):
  - Ambulatorium Barbara Bazela, Elblag, Warminsko-Mazurki
  - NZOZ ZDROWIE Osteo-Medic, Bialystok
  - Poradnia Diabetologiczna SN ZOZ Lege Artis, Bialystok
  - NZOZ Diab-Endo-Met, Krakow
  - Gabinet Lekarski Malgorzata Saryusz-Wolska, Lodz
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska S.K.A., Lodz
  - NZOZ Przychodnia Specjalistyczna MEDICA, Lublin
  - NZOZ Przychodnia Specjalistyczna Henryk RudzkiAndrzej Wittek, Ruda Śląska
- Puerto Rico (3):
  - Latin Clinical Trial Center, San Juan, PR
  - GCM Medical Group PSC, San Juan, PR
  - San Miguel Medical, Trujillo Alto, PR
- Romania (10):
  - S. C. Grandmed S.R.L., Str., Oradea, Bihor County
  - SC Diamed Obesity SRL, Galati, Galați County
  - Spitalul Judetean de Urgenta Satu Mare, Satu Mare, Jud Satu-Mare
  - CMI DNBM Dr. Pop Lavinia, Baia Mare, Maramureş
  - Cosamext SRL, Târgu Mureş, Mureș County
  - Societatea Civila Medicala "Dr. Paveliu", Bucharest, Sect.5
  - Centrul Medical de Diagnostic si Tratament Ambulatoriu Neomed SRL, Brasov
  - Cabinetul Medical Nicodiab SRL, Bucharest
  - SC Nutrilife SRL, Bucharest
  - Consultmed SRL, Iași
- South Korea (10):
  - Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggido
  - Seoul St. Mary's Hospital, Seoul, Korea
  - Korea University Ansan Hospital, Ansan-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Kyunghee University Hospital at Gangdong, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hospital Infanta Luisa, Seville, Andalusia
  - Hospital Universitario Marques De Valdecilla, Santander, Cantabria
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcón, Madrid
  - Instituto de Ciencias médicas, Alicante
  - Hospital Clinico Universitario San Cecilio, Granada
  - Clinica Juaneda, Palma de Mallorca
  - Clinica Nuevas Tecnologias en Diabetes y Endocrinologia, Seville
  - Policlinica Galileo, Teruel
- Taiwan (9):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung City
  - Taipei Medical University- Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Kuang Tien General Hospital, Taichung County
  - National Cheng Kung University Hospital, Tainan
  - Chi-Mei Medical Center, Tainan
  - Taipei Veterans General Hospital, Taipei
- Ukraine (4):
  - Dnipro City Clinical Hospital #9, Dnipro
  - V.P. Komisarenko Institute of Endocrinology and Metabolism of NAMS of Ukraine, Kyiv
  - Communal Institution "Poltava Reg.Cl.H. n.a.M.V.Sklifosovskogo", Poltava
  - Vinnytsia Regional Clinical Highly Specialized Endocrinology Center, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Sattar N, Neeland IJ, Dahlqvist Leinhard O, Fernandez Lando L, Bray R, Linge J, Rodriguez A. Tirzepatide and muscle composition changes in people with type 2 diabetes (SURPASS-3 MRI): a post-hoc analysis of a randomised, open-label, parallel-group, phase 3 trial. Lancet Diabetes Endocrinol. 2025 Jun;13(6):482-493. doi: 10.1016/S2213-8587(25)00027-0. Epub 2025 Apr 30. PMID 40318682
- [Derived] De Block C, Peleshok J, Wilding JPH, Kwan AYM, Rasouli N, Maldonado JM, Wysham C, Liu M, Aleppo G, Benneyworth BD. Post Hoc Analysis of SURPASS-1 to -5: Efficacy and Safety of Tirzepatide in Adults with Type 2 Diabetes are Independent of Baseline Characteristics. Diabetes Ther. 2025 Jan;16(1):43-71. doi: 10.1007/s13300-024-01660-0. Epub 2024 Nov 12. PMID 39531161
- [Derived] Boye KS, Sapin H, Dong W, Williamson S, Lee CJ, Thieu VT. Improved Glycaemic and Weight Management Are Associated with Better Quality of Life in People with Type 2 Diabetes Treated with Tirzepatide. Diabetes Ther. 2023 Nov;14(11):1867-1887. doi: 10.1007/s13300-023-01457-7. Epub 2023 Sep 5. PMID 37668888
- [Derived] Boye KS, Thieu VT, Sapin H, Lee CJ, Lando LF, Brown K, Bray R, Wiese RJ, Patel H, Rodriguez A, Yu M. Patient-Reported Outcomes in People with Type 2 Diabetes Receiving Tirzepatide in the SURPASS Clinical Trial Programme. Diabetes Ther. 2023 Nov;14(11):1833-1852. doi: 10.1007/s13300-023-01451-z. Epub 2023 Aug 1. PMID 37526908
- [Derived] Viljoen A, Pantalone KM, Galindo RJ, Cui X, Huh R, Hemmingway A, Fernandez Lando L, Patel H. Time to Reach Glycaemic and Body Weight Loss Thresholds with Tirzepatide in Patients with Type 2 Diabetes: A Pre-planned Exploratory Analysis of SURPASS-2 and SURPASS-3. Diabetes Ther. 2023 May;14(5):925-936. doi: 10.1007/s13300-023-01398-1. Epub 2023 Mar 31. PMID 37000390
- [Derived] Gastaldelli A, Cusi K, Fernandez Lando L, Bray R, Brouwers B, Rodriguez A. Effect of tirzepatide versus insulin degludec on liver fat content and abdominal adipose tissue in people with type 2 diabetes (SURPASS-3 MRI): a substudy of the randomised, open-label, parallel-group, phase 3 SURPASS-3 trial. Lancet Diabetes Endocrinol. 2022 Jun;10(6):393-406. doi: 10.1016/S2213-8587(22)00070-5. Epub 2022 Apr 22. PMID 35468325
- [Derived] Battelino T, Bergenstal RM, Rodriguez A, Fernandez Lando L, Bray R, Tong Z, Brown K. Efficacy of once-weekly tirzepatide versus once-daily insulin degludec on glycaemic control measured by continuous glucose monitoring in adults with type 2 diabetes (SURPASS-3 CGM): a substudy of the randomised, open-label, parallel-group, phase 3 SURPASS-3 trial. Lancet Diabetes Endocrinol. 2022 Jun;10(6):407-417. doi: 10.1016/S2213-8587(22)00077-8. Epub 2022 Apr 22. PMID 35468321
- [Derived] Sattar N, McGuire DK, Pavo I, Weerakkody GJ, Nishiyama H, Wiese RJ, Zoungas S. Tirzepatide cardiovascular event risk assessment: a pre-specified meta-analysis. Nat Med. 2022 Mar;28(3):591-598. doi: 10.1038/s41591-022-01707-4. Epub 2022 Feb 24. PMID 35210595
- [Derived] Ludvik B, Giorgino F, Jodar E, Frias JP, Fernandez Lando L, Brown K, Bray R, Rodriguez A. Once-weekly tirzepatide versus once-daily insulin degludec as add-on to metformin with or without SGLT2 inhibitors in patients with type 2 diabetes (SURPASS-3): a randomised, open-label, parallel-group, phase 3 trial. Lancet. 2021 Aug 14;398(10300):583-598. doi: 10.1016/S0140-6736(21)01443-4. Epub 2021 Aug 6. PMID 34370970
- See also: A Study of Tirzepatide (LY3298176) Versus Insulin Degludec in Participants With Type 2 Diabetes — https://trials.lillytrialguide.com/en-US/trial/76cf8Mdt50agkx23op5368

RESULTS

PARTICIPANT FLOW:
Groups:
- 15 mg Tirzepatide: 15 mg tirzepatide administered SC once a week SC.
- Insulin Degludec: Insulin degludec administered SC once a day. Doses were individualized and titrated according to protocol-defined targets.
  The starting dose of insulin degludec was 10 IU/day ideally at bedtime, titrated to a fasting blood glucose (FBG) <90 milligram per Deciliter (mg/dL), following a treat-to-target (TTT) algorithm based on the last 3 FBG values.
Period: Overall Study
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Degludec
Started | 359 | 361 | 359 | 365
Received at Least One Dose of Study Drug | 358 | 360 | 359 | 360
Completed | 333 | 321 | 340 | 331
Not Completed | 26 | 40 | 19 | 34
Not completed — Adverse Event | 5 | 7 | 3 | 1
Not completed — Death | 1 | 2 | 1 | 1
Not completed — Lost to Follow-up | 8 | 9 | 5 | 5
Not completed — Physician Decision | 0 | 2 | 2 | 2
Not completed — Protocol Violation | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 17 | 7 | 22
Not completed — Personal Reason | 2 | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Degludec | Total
Number analyzed (Participants) | 359 | 361 | 359 | 365 | 1444
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.20 (10.13) | 57.40 (9.66) | 57.50 (10.24) | 57.50 (10.08) | 57.40 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 158 | 165 | 165 | 148 | 636
  Male | 201 | 196 | 194 | 217 | 808
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 109 | 108 | 96 | 108 | 421
  Not Hispanic or Latino | 247 | 253 | 259 | 256 | 1015
  Unknown or Not Reported | 3 | 0 | 4 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2 | 4
  Asian | 20 | 19 | 20 | 19 | 78
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 2 | 1 | 4
  Black or African American | 13 | 12 | 8 | 11 | 44
  White | 324 | 329 | 327 | 332 | 1312
  More than one race | 1 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 57 | 54 | 56 | 57 | 224
  Austria | 7 | 8 | 4 | 8 | 27
  Greece | 33 | 35 | 35 | 34 | 137
  Hungary | 36 | 37 | 37 | 37 | 147
  Italy | 6 | 8 | 8 | 8 | 30
  Poland | 33 | 33 | 33 | 33 | 132
  Puerto Rico | 8 | 7 | 11 | 9 | 35
  Romania | 54 | 54 | 53 | 53 | 214
  South Korea | 9 | 10 | 8 | 9 | 36
  Spain | 21 | 21 | 22 | 22 | 86
  Taiwan | 9 | 8 | 10 | 9 | 36
  Ukraine | 11 | 11 | 12 | 11 | 45
  United States | 75 | 75 | 70 | 75 | 295
Hemoglobin A1c [Mean (Standard Deviation); unit: Percentage of HbA1c] — Population: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Hemoglobin A1c Analysis Population Description: All randomized participants who had a HbA1c baseline value.
  Percentage of HbA1c
    number analyzed (Participants) | 358 | 360 | 359 | 360 | 1437
    (all) | 8.17 (0.89) | 8.18 (0.89) | 8.21 (0.94) | 8.12 (0.94) | 8.17 (0.91)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c) (10 mg and 15 mg)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with covariates Baseline + Pooled Country + Baseline Oral Antihyperglycemic Medication (OAM) Use (Metformin (Met), Met plus SGLT-2i) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: All randomized participants who received at least one dose of study drug and had a baseline and at least 1 post-baseline value, excluding participants discontinuing study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or stopping study drug (last dose date +7 days)
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Degludec
Number analyzed (Participants) | 291 | 294 | 317
Percentage of HbA1c | -2.20 (0.051) | -2.37 (0.050) | -1.34 (0.049)
Statistical Analysis 1: Comparison: 10 mg Tirzepatide vs Insulin Degludec; Test type: Non-Inferiority — The study was powered for superiority in HbA1c. The sample size provided >99% power to show noninferiority assuming a 0.3% NI boundary, 0.35% greater mean reduction in tirzepatide doses compared to insulin degludec, 1:1:1:1 randomization, a common SD of 1.1%, 1 sided significance level of 0.0125, and a dropout rate of 28%; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.86, 95% CI 2-sided [-1.00 to -0.72]
Statistical Analysis 2: Comparison: 15 mg Tirzepatide vs Insulin Degludec; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; LS Mean Difference = -1.04, 95% CI 2-sided [-1.17 to -0.90]

2. Secondary Outcome: Change From Baseline in HbA1c (5 mg)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least Squares (LS) mean was determined by mixed-model repeated measures (MMRM) model with covariates Baseline + Pooled Country + Baseline OAM Use (Met, Met plus SGLT-2i) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | 5 mg Tirzepatide | Insulin Degludec
Number analyzed (Participants) | 312 | 317
Percentage of HbA1c | -1.93 (0.050) | -1.34 (0.049)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Degludec; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Mixed Models Analysis; LS Mean Difference = -0.59, 95% CI 2-sided [-0.73 to -0.45]

3. Secondary Outcome: Change From Baseline in Body Weight
Description: LS mean was determined by MMRM model with Baseline + Pooled Country + Baseline OAM Use (Met, Met plus SGLT-2i) + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment + Time + Treatment*Time (Type III sum of squares) as covariates.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kilograms (kg)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Degludec
Number analyzed (Participants) | 310 | 291 | 295 | 317
Kilograms (kg) | -7.5 (0.37) | -10.7 (0.37) | -12.9 (0.37) | 2.3 (0.37)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Degludec; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -9.8, 95% CI 2-sided [-10.8 to -8.8]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Degludec; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -13.0, 95% CI 2-sided [-14.0 to -11.9]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Degludec; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean Difference = -15.2, 95% CI 2-sided [-16.2 to -14.2]

4. Secondary Outcome: Change From Baseline in Fasting Serum Glucose
Description: LS mean was determined by MMRM model with variables Baseline + Pooled Country + Baseline OAM Use (Met, Met plus SGLT-2i) + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligram per Deciliter (mg/dL)
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Degludec
Number analyzed (Participants) | 309 | 291 | 293 | 314
milligram per Deciliter (mg/dL) | -48.2 (1.82) | -54.8 (1.86) | -59.2 (1.85) | -55.7 (1.81)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Degludec; Test type: Superiority; p = 0.004, Mixed Models Analysis; LS Mean Difference = 7.5, 95% CI 2-sided [2.4 to 12.5]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Degludec; Test type: Superiority; p = 0.751, Mixed Models Analysis; LS Mean Difference = 0.8, 95% CI 2-sided [-4.3 to 5.9]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Degludec; Test type: Superiority; p = 0.168, Mixed Models Analysis; LS Mean Difference = -3.6, 95% CI 2-sided [-8.7 to 1.5]

5. Secondary Outcome: Percentage of Participants Achieving an HbA1c Target Value of <7%
Description: Hemoglobin A1c (HbA1c) is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. Imputed data includes observed value and imputed value if endpoint measure is missing. Missing endpoint measures are imputed by predictions from an MMRM analysis model using observed data in the efficacy analysis set and adjusted for Baseline Value, Pooled Country, Baseline OAM Use (Met, Met plus SGLT-2i), Treatment, Visit and Visit*Treatment.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Degludec
Number analyzed (Participants) | 353 | 350 | 353 | 351
percentage of participants | 82.44 | 89.71 | 92.63 | 61.25
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Degludec; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 3.45, 95% CI 2-sided [2.38 to 5.01]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Degludec; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 7.02, 95% CI 2-sided [4.55 to 10.84]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Degludec; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 10.79, 95% CI 2-sided [6.65 to 17.48]

6. Secondary Outcome: Mean Change From Baseline in Daily Average 7-Point Self-Monitored Blood Glucose (SMBG) Values
Description: The self-monitored plasma glucose (SMBG) data were collected at the following 7 time points: Morning Premeal - Fasting, Morning 2-hour Postmeal, Midday Premeal, Midday 2-hour Postmeal, Evening Premeal, Evening 2-hour Postmeal and Bedtime. LS mean was determined by mixed-model repeated measures (MMRM) model with variables Baseline + Baseline HbA1c Group (<=8.5%, >8.5%) + Pooled Country + Baseline OAM Use (Met, Met plus SGLT-2i) + Treatment + Time + Treatment*Time (Type III sum of squares).
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Degludec
Number analyzed (Participants) | 281 | 263 | 274 | 288
mg/dL | -52.6 (1.20) | -59.7 (1.22) | -60.6 (1.20) | -48.0 (1.18)

7. Secondary Outcome: Percentage of Participants Who Achieved Weight Loss ≥5%
Description: Percentage of Participants who Achieved Weight Loss ≥5%
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Degludec
Number analyzed (Participants) | 353 | 350 | 353 | 351
percentage of participants | 66.01 | 83.71 | 87.82 | 6.27
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Degludec; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 29.78, 95% CI 2-sided [18.35 to 48.35]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Degludec; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 79.88, 95% CI 2-sided [47.56 to 134.17]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Degludec; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 110.77, 95% CI 2-sided [64.73 to 189.55]

8. Secondary Outcome: Diabetes Treatment Satisfaction as Measured by the Diabetes Treatment Satisfaction Questionnaire, Change Version (DTSQc) Hyperglycemia, Hypoglycemia and Treatment Satisfaction Score
Description: DTSQc, an 8-item questionnaire, assesses relative change in treatment satisfaction perceived frequency of hyperglycemia, and perceived frequency of hypoglycemia from baseline to week 52 or early termination.The treatment satisfaction score ranges from -18 to 18 where the higher the score the greater the improvement in satisfaction with treatment. The lower the score the greater the deterioration in satisfaction with treatment. The hyperglycemia and hypoglycemia scores range from -3 to 3 where negative scores indicate fewer problems with blood glucose levels and positive scores indicate more problems than before. LS mean was determined by ANCOVA model for endpoint measures: Variable = Baseline DTSQs + Pooled Country + Baseline HbA1c Group (<=8.5%, >8.5%) + Baseline OAM Use (Met, Met plus SGLT-2i) + Treatment (Type III sum of squares).
Time Frame: Week 52
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Degludec
Number analyzed (Participants) | 306 | 293 | 292 | 313
units on a scale
  Hyperglycemia: number analyzed (Participants) | 306 | 293 | 292 | 312
  Hyperglycemia | -1.4 (0.11) | -1.4 (0.11) | -1.6 (0.11) | -1.1 (0.11)
  Hypoglycemia | -1.1 (0.12) | -0.9 (0.12) | -1.0 (0.12) | -0.7 (0.12)
  Treatment Satisfaction Score: number analyzed (Participants) | 305 | 293 | 292 | 313
  Treatment Satisfaction Score | 15.6 (0.27) | 15.5 (0.28) | 15.6 (0.28) | 12.6 (0.27)
Statistical Analysis 1: Comparison: 5 mg Tirzepatide vs Insulin Degludec; Hyperglycemia; Test type: Superiority; p = 0.096, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-0.57 to 0.05]
Statistical Analysis 2: Comparison: 10 mg Tirzepatide vs Insulin Degludec; Hyperglycemia; Test type: Superiority; p = 0.113, ANCOVA; LS Mean Difference = -0.25, 95% CI 2-sided [-0.57 to 0.06]
Statistical Analysis 3: Comparison: 15 mg Tirzepatide vs Insulin Degludec; Hyperglycemia; Test type: Superiority; p = 0.003, ANCOVA; LS Mean Difference = -0.47, 95% CI 2-sided [-0.78 to -0.16]
Statistical Analysis 4: Comparison: 5 mg Tirzepatide vs Insulin Degludec; Hypoglycemia; Test type: Superiority; p = 0.014, ANCOVA; LS Mean Difference = -0.41, 95% CI 2-sided [-0.74 to -0.08]
Statistical Analysis 5: Comparison: 10 mg Tirzepatide vs Insulin Degludec; Hypoglycemia; Test type: Superiority; p = 0.280, ANCOVA; LS Mean Difference = -0.18, 95% CI 2-sided [-0.51 to 0.15]
Statistical Analysis 6: Comparison: 15 mg Tirzepatide vs Insulin Degludec; Hypoglycemia; Test type: Superiority; p = 0.129, ANCOVA; LS Mean Difference = -0.26, 95% CI 2-sided [-0.59 to 0.07]
Statistical Analysis 7: Comparison: 5 mg Tirzepatide vs Insulin Degludec; Treatment Satisfaction Score; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 3.01, 95% CI 2-sided [2.26 to 3.75]
Statistical Analysis 8: Comparison: 10 mg Tirzepatide vs Insulin Degludec; Treatment Satisfaction Score; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 2.90, 95% CI 2-sided [2.15 to 3.65]
Statistical Analysis 9: Comparison: 15 mg Tirzepatide vs Insulin Degludec; Treatment Satisfaction Score; Test type: Superiority; p < 0.001, ANCOVA; LS Mean Difference = 2.99, 95% CI 2-sided [2.24 to 3.74]

9. Secondary Outcome: Rate of Hypoglycemia With Blood Glucose <54 Milligram/Deciliter (mg/dL) [<3.0 (Millimole/Liter (mmol/L))] or Severe Hypoglycemia
Description: The hypoglycemia events were defined by participant reported events with blood glucose <54mg/dL (<3.0 mmol/L) or severe hypoglycemia. Severe hypoglycemia is defined as an episode with severe cognitive impairment requiring the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. These episodes may be associated with sufficient neuroglycopenia to induce seizure or coma. The rate of postbaseline hypoglycemia was estimated by negative binomial model: Number of episodes = Pooled Country + Baseline OAM Use (Met, Met plus SGLT-2i) + Baseline HbA1c Group (<=8.5%, >8.5%) + Treatment, with log (exposure in days/365.25) as an offset variable.
Time Frame: Baseline through Safety Follow-Up (Up to Week 56)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Episodes/participant/365.25 days
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Degludec
Number analyzed (Participants) | 356 | 360 | 359 | 358
Episodes/participant/365.25 days | 0.0137 (0.0056) | 0.0108 (0.0044) | 0.0275 (0.0143) | 0.1020 (0.0568)

ADVERSE EVENTS:
Time Frame: Baseline Up To 56 Weeks
Description: All participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- 10 mg Tirzepatide: 5 milligrams (mg) tirzepatide administered subcutaneously (SC) once a week.
Arm/Group | 5 mg Tirzepatide | 10 mg Tirzepatide | 15 mg Tirzepatide | Insulin Degludec
All-Cause Mortality (participants affected / at risk) | 1/358 | 2/360 | 1/359 | 1/360
Serious Adverse Events (participants affected / at risk) | 29/358 | 20/360 | 26/359 | 22/360
Other Adverse Events (participants affected / at risk) | 124/358 | 157/360 | 179/359 | 66/360
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 5 mg Tirzepatide (N=358) | 10 mg Tirzepatide (N=360) | 15 mg Tirzepatide (N=359) | Insulin Degludec (N=360)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Arrhythmogenic right ventricular dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis alcoholic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Segmental diverticular colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Necrosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Malignant biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis orbital (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hepatitis e (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0/158 (0) | 1/165 (1) | 0/165 (0) | 0/147 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sars-cov-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma stage iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/200 (1) | 0/195 (0) | 0/194 (0) | 0/213 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/158 (0) | 1/165 (1) | 0/165 (0) | 0/147 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression suicidal (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0/158 (0) | 0/165 (0) | 1/165 (1) | 0/147 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5 mg Tirzepatide (N=358) | 10 mg Tirzepatide (N=360) | 15 mg Tirzepatide (N=359) | Insulin Degludec (N=360)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 17 (28) | 23 (46) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 55 (92) | 59 (97) | 56 (107) | 14 (18)
Dyspepsia (Gastrointestinal disorders) | 14 (14) | 32 (39) | 18 (28) | 0 (0)
Nausea (Gastrointestinal disorders) | 41 (86) | 81 (140) | 85 (240) | 6 (6)
Vomiting (Gastrointestinal disorders) | 21 (29) | 34 (53) | 36 (63) | 4 (4)
Nasopharyngitis (Infections and infestations) | 11 (11) | 14 (15) | 15 (16) | 22 (27)
Lipase increased (Investigations) | 21 (25) | 16 (18) | 20 (21) | 7 (7)
Decreased appetite (Metabolism and nutrition disorders) | 22 (23) | 37 (59) | 43 (54) | 2 (2)
Hypertension (Vascular disorders) | 11 (11) | 7 (8) | 11 (11) | 21 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT03882970/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/70/NCT03882970/SAP_001.pdf